CLINICAL TRIAL: NCT01429337
Title: An Open-label, Parallel Group, Phase I Study to Assess the Pharmacokinetics and Safety of Midostaurin in Subjects With Impaired Hepatic Function and Subjects With Normal Hepatic Function.
Brief Title: PK and Safety of Midostaurin in Subjects With Impaired Hepatic Function and Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CPKC412A2116; 2010-020694-16 (EudraCT Number)
Record Dates: First submitted 2011-07-12; First posted 2011-09-07 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Hepatic Impairment
Keywords: Pharmacokinetics; Hepatic impaired patients; Healthy volunteers; Varying degrees of hepatic impairment
MeSH Terms: interventions — midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Normal hepatic function - group 1 (Experimental): Matched control for group 2 and 3 - healthy volunteers matched with respect to age, body weight, BMI and gender to subjects in mild and moderate hepatic function groups. Subjects will be treated with midostaurin 50mg b.i.d from days 1-6 and 50mg o.d on day 7.
  Interventions: Drug: Midostaurin
- Mild hepatic impairment - group 2 (Experimental): Subjects with mild impaired hepatic function - Child Pugh A classification score 5-6. Subjects will be treated with midostaurin 50mg b.i.d from days 1-6 and 50mg o.d on day 7.
  Interventions: Drug: Midostaurin
- Moderate hepatic impairment - group 3 (Experimental): Subjects with moderate hepatic function - Child Pugh B classification score 7-9. Subjects will be treated with midostaurin 50mg b.i.d from days 1-6 and 50mg o.d on day 7.
  Interventions: Drug: Midostaurin
- Severe hepatic impairment - group 4 (Experimental): Subjects with severe hepatic impairment function - Child Pugh C classification score 10-15. Subjects will be treated with a single dose of midostaurin of 50mg on day 1.
  Interventions: Drug: Midostaurin
- Normal hepatic function - group 5 (Experimental): Matched control for group 4 - healthy volunteers matched with respect to age, body weight, BMI and gender to subjects in severe hepatic function group. Subjects will be treated with a single dose of midostaurin of 50mg on day 1.
  Interventions: Drug: Midostaurin

INTERVENTIONS:
Drug: Midostaurin — Midostaurin 25 mg soft gelatin capsules (2 capsules). The midostaurin capsules will be administered orally with 240 mL of non-carbonated water in the morning (between 8-10 AM), and in the evening (after a 12 hour break) from Day 1 to Day 6. On Day 7, midostaurin will be administered in the morning only (between 8-10 AM).
  Other Names: PKC412
  Arms: Mild hepatic impairment - group 2; Moderate hepatic impairment - group 3; Normal hepatic function - group 1
Drug: Midostaurin — Midostaurin 25 mg soft gelatin capsules (2 capsules). The midostaurin capsules will be administered orally with 240 mL of non-carbonated water in the morning (between 8-10 AM) on Day 1 only.
  Other Names: PKC412
  Arms: Normal hepatic function - group 5; Severe hepatic impairment - group 4

SUMMARY:
The purpose of this international study was to assess the effect of varying degrees of impaired hepatic function compared to a normal hepatic function (Child-Pugh classification) on the pharmacokinetics and safety of midostaurin.

DETAILED DESCRIPTION:
Midostaurin was developed for the treatment of patients with hematological and nonhematological malignancies. However, disease complications and various co-medications made it difficult to perform a hepatic impairment study in the targeted patient population.

Metabolism and elimination of midostaurin predominantly occurs in the liver. Patients with impaired hepatic function may have a higher risk to have a decreased elimination or metabolism of midostaurin which may lead to increased systemic exposure or toxicity, hence understanding the impact of an impaired hepatic function on midostaurin PK is important.

Cumulative safety data from over 900 subjects exposed to midostaurin showed that the drug was well tolerated in patients and in healthy subjects, thus, it was appropriate and justifiable to study midostaurin in subjects with varying degrees of hepatic impairment.

Due to the difficulty in enrolling subjects with severe hepatic impairment, an interim analysis was performed when all mild and moderate hepatic impaired subjects, and the respective control subjects, had completed the trial, in order to obtain interim results on the PK and safety of midostaurin in patients with mild and moderate hepatic impairment. The protocol was amended in April 2018 to make the inclusion / exclusion criteria more fitting with enrolling the severe hepatic impairment group. The final study analysis was performed when all severe hepatic impaired subjects, and the matching controls, had completed the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult male or female subjects age 18-70 years
* Negative serum beta-hCG pregnancy test for all women prior to starting treatment
* Normal vital signs, body weight, BMI and laboratory test results
* Willing to comply with dietary, fluid and lifestyle restrictions
* Able to communicate well with the Investigator and comply with the requirements of the study.

Additional Inclusion Criteria for hepatic impaired subjects

* Physical signs consistent with hepatic impairment
* CPC score consistent with degree of hepatic impairment
* Serum creatinine <=2xULN
* ANC >1000cells/mm3, hemaglobin >9g/dL, platelet count > 50,000/mm3 (group 2-3 only)

Key Exclusion Criteria:

* Significant neurologic or psychiatric disorder which could compromise participation in the study.
* History of: seizures requiring anti-convulsant therapy; unstable COPD; GI or rectal bleeding 3 weeks prior to study start; Myocardial Infarction within 12 months; unstable or poorly controlled angina or other clinically significant heart disease; clinically significant urinary obstruction or difficulty voiding; clinically significant ECG abnormalities or long QT-interval syndrome; pancreatic injury or pancreatitis
* Concurrent severe / uncontrolled medical conditions
* Significant illness within 2 weeks prior to dosing or hospitalisation within 4 weeks prior to dosing
* Any surgical or medical condition that may significantly affect absorption, distribution, metabolism or excretion of drugs
* Clinically significant ECG abnormalities at screening
* Cotinine levels greater than 500ng/mL (group 1-3) or smokers not willing to limit tobacco or nicotine products equivalent to 10 cigarettes per day (group 4 and 5) for 1 week prior to dosing and throughout hospital confinement
* Consumption of alcohol within 3 days (group 1-3) or within 2 days (groups 4 and 5) prior to dosing or during the study.
* Administration of CYP3A4/5 or P-gp inducing or inhibiting drugs within 14 days prior to dosing or during the study
* Sexually active males unless they use condom during intercourse while taking midostaurin and for at least 3 months after the last exposure to drug.
* Use of any prescription drug within 2 weeks or over the counter medication within 72 hours prior to dosing
* Consumption of grapefruit, grapefruit juice, Seville oranges, start fruit / juice within 72 hours prior to dosing

Additional exclusion criteria for healthy controls

* Clinical evidence of liver disease or liver injury
* Positive HBsAg or Hep C test result

Additional exclusion criteria for hepatic impairment subjects

* Symptoms or history of >=G3 hepatic encephalopathy; surgical portosystemic shunt
* PTT >2.5xULN; INR >3; Total bilirubin >6mg/dL
* Evidence of progressive liver disease within 4 weeks prior to starting study
* Clinical evidence of severe >=G3 ascites (groups 2 and 3)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-03-07 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-05-09 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentrations (Cmax) for midostaurin and its metabolites, CGP52421 and CGP62221 | at different timepoints from Day 1 to Day 7
  In subjects with Child Pugh A, Child Pugh B (and matching healthy volunteers) Cmax will be measured at Day 1 and Day 7. In subjects with Child Pugh C (and matching healthy volunteers) Cmax will be measured at Day 1

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (AEs) | During the study and until 28 days follow-up period
  Safety and tolerability of midostaurin measured by the number of treatment emergent adverse events in subjects with hepatic impairment (and matching healthy volunteers)
CYP3A4 induction by midostaurin in the hepatic impaired population | At different timepoints from Day 3 to Day 11
  CYP3A4 induction will be measured by assessing endogenous biomarkers (6beta-hydroxycortisol to cortisol ratio) applicable to multiple dosing Child Pugh A and Child Pugh B subjects and matching healthy volunteers)
Protein binding (free fraction) of midostaurin and it's metabolites | Day 1 and Day 7
  Free fraction of midostaurin and it's metabolites, CGP62221 and CGP52421, will be assessed by measuring their unbound concentration in plasma samples 3 hours post last dose on Day 1 (group 4 and 5) and Day 7 (group 1-3).
Apparent volume of distribution (Vz/F) of midostaurin | Day 1 and Day 7
  In subjects with Child Pugh A and Child Pugh B (and matching healthy volunteers), volume of distribution will be measured on Day 7. In subjects with Child Pugh C (and healthy volunteers), volume of distribution will be measured at Day 1.
Total body apparent clearance of drug (CL/F) of midostaurin | Day 1 and Day 7
  In subjects with Child Pugh A and Child Pugh B (and matching healthy volunteers), total body clearance will be measured on Day 7. In subjects with Child Pugh C (and healthy volunteers), total body clearance will be measured at Day 1.
Elimination half life (t½) of midostaurin and its metabolites, CGP52421 and CGP62221 | Day 1 and Day 7
  In subjects with Child Pugh A and Child Pugh B (and matching healthy volunteers), elimination half life will be measured on Day 7. In subjects with Child Pugh C (and healthy volunteers), elimination half life will be measured at Day 1.
Time to maximum plasma concentration (tmax) for midostaurin and its metabolites, CGP52421 and CGP62221 | Day 1 and Day 7
  In subjects with Child Pugh A and Child Pugh B (and matching healthy volunteers), tmax will be measured at Day 1 and Day 7. In subjects with Child Pugh C (and healthy volunteers), tmax will be measured at Day 1.
Area under the plasma concentration versus time curves (AUCs) for midostaurin and its metabolites, CGP52421 and CGP62221 | Day 1 and Day 7
  In subjects with Child Pugh A and Child Pugh B (and matching healthy volunteers), AUC will be measured at Day 1 and Day 7. In subjects with Child Pugh C (and healthy volunteers), AUC will be measured at Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- American Research Corporation Inc, San Antonio, Texas, United States
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Sofia, Bulgaria
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
- Novartis Investigative Site, Kaunas, LTU, Lithuania
- Novartis Investigative Site, Cluj-Napoca, Napoca, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Novartis clinical trials results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17823